CLINICAL TRIAL: NCT01441336
Title: Laparoscopic Gastrectomy for Advanced Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyung-Ho Kim, Principal Investigator, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUBHGS02
Record Dates: First submitted 2011-09-25; First posted 2011-09-27 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Advanced Gastric Cancer; Laparoscopic Gastrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Laparoscopic gastrectomy (Experimental): Laparoscopic gastrectomy procedure:
  D2 lymphadenectomy & total omentectomy in case of tumor with serosa exposure under laparoscopic exploration
  Interventions: Procedure: Laparoscopic gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic gastrectomy — Operative procedure: laparoscopic gastrectomy(D2 lymphadenectomy according to JGCA guideline and total omentectomy for tumor with serosa exposure)

SUMMARY:
Although laparoscopic gastrectomy (LG) is widely used for the treatment of early gastric cancer, there have been few reports of the efficacy of LAG in the management of advanced gastric cancer(AGC). The aim of this study is to evaluate the surgical outcomes and oncologic safety of laparoscopic gastrectomy for AGC.

DETAILED DESCRIPTION:
Prospective phase II clinical trial to evaluate technical and oncological safety of LG for AGC

LG procedure for AGC:

D2 lymphadenectomy Total omentectomy for tumor with serosa exposure under laparoscopic exploration

Primary end point: 3 year disease free survival secondary end point: postoperative outcomes, morbidity and mortality, 3,5 and 7 year overall survival, Quality of life, recurrence pattern

Study duration: 7 years(enrollment: 4year, follow-up: 3year)

ELIGIBILITY:
Inclusion Criteria:

* Age 20-80
* informed consent
* no other malignancies
* cT2N0-cT3N2 according to JGCA 2nd edition
* ASA score<3

Exclusion Criteria:

* distant metastasis(P1 or M1) under laparoscopic exploration
* Conglomerated N2
* early gastric cancer in permanent pathologic report

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2008-11; Primary Completion 2012-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
3 year recurrence free survival | Postoperative 3 year
  Evaluation of recurrence after regular 3 months follow-up using tumor marker, chest x-ray, endoscopy and computed tomograhy.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang L, Hong H, Zang L, Dong F, Lu A, Feng B, He Z, Xue P, Cai Z, Zheng M, Ma J. Application Value of 4K High-Definition System in Laparoscopic Gastrectomy: Preliminary Results and Initial Experience. J Laparoendosc Adv Surg Tech A. 2022 Feb;32(2):137-141. doi: 10.1089/lap.2020.0931. Epub 2021 May 7. PMID 33970027
- [Derived] Ahn SH, Kang SH, Lee Y, Min SH, Park YS, Park DJ, Kim HH. Long-term Survival Outcomes of Laparoscopic Gastrectomy for Advanced Gastric Cancer: Five-year Results of a Phase II Prospective Clinical Trial. J Gastric Cancer. 2019 Mar;19(1):102-110. doi: 10.5230/jgc.2019.19.e6. Epub 2019 Mar 12. PMID 30944763
- [Derived] Lee JH, Son SY, Lee CM, Ahn SH, Park DJ, Kim HH. Morbidity and mortality after laparoscopic gastrectomy for advanced gastric cancer: results of a phase II clinical trial. Surg Endosc. 2013 Aug;27(8):2877-85. doi: 10.1007/s00464-013-2848-0. Epub 2013 Feb 13. PMID 23404155